CLINICAL TRIAL: NCT06971211
Title: An Open, Single Arm, Multicenter Clinical Study on the First-line Treatment of Metastatic Castration Resistant Prostate Cancer With Radiotherapy Combined With Fuzuloparib and Abiraterone Acetate Tablets（Ⅱ）
Brief Title: Radiotherapy Combined With Fluzopanib and Abiraterone Acetate Tablets (II) Treatment for mCRPC
Acronym: PARTOM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jianbin Bi (Other)
Responsible Party: Sponsor-Investigator, Jianbin Bi, Investigator, First Hospital of China Medical University
Organization: First Hospital of China Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FirstHCMU-JBi-PARTOM
Record Dates: First submitted 2025-04-18; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: prostate cancer; fuzuloparib; abiraterone acetate; Intensity modulated radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated; fluzoparib; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): Induction therapy,patients were treated with intensity-modulated radiation therapy (IMRT) combined with fluzoparib,abiraterone acetate tablets (II), and prednisone. Maintenance treatment,patients received the same doses of fluzoparib,abiraterone acetate (II), and prednisone. Each treatment cycle lasted 28 days.
  Interventions: Drug: Intensity-modulated radiation therapy (IMRT) in combination with fluzoparib, abiraterone acetate tablets (II), and prednisone.

INTERVENTIONS:
Drug: Intensity-modulated radiation therapy (IMRT) in combination with fluzoparib, abiraterone acetate tablets (II), and prednisone. — Induction therapy, fluzoparib (150mg BID orally), abiraterone acetate tablets (II) (300mg QD orally), and prednisone (5mg BID orally). IMRT was administered as follows: For patients with low metastatic burden tumors: Prostate ± pelvic lymph node radiation + metastatic lesion radiation.For patients with non-low metastatic burden tumors: Prostate±pelvic lymph node radiation.IMRT dosage:Prostate: 70 Gy in 28 fractions (2.5 Gy/fraction, 5 fractions per week).Pelvic lymph nodes: 50.4 Gy in 28 fractions (1.8 Gy/fraction, 5 fractions per week).Fluzoparib and abiraterone acetate (II) were administered concurrently with radiotherapy. Maintenance treatment,patients received the same doses of fluzoparib,abiraterone acetate (II), and prednisone. Each treatment cycle lasted 28 days.
  Other Names: Treatment group

SUMMARY:
This study is an open label, single arm, multicenter clinical trial. The aim of this study is to evaluate the efficacy, safety, and quality of life of radiotherapy combined with Fuzuloparib and Abiraterone Acetate Tablets（Ⅱ） as first-line treatment for castration resistant prostate cancer patients. The study aims to enroll 40 eligible subjects with PSA response rate (PSA 50) as the primary endpoint.

DETAILED DESCRIPTION:
This study is an open-label, single-arm, multicenter clinical trial designed to evaluate the efficacy, safety, and quality of life of first-line treatment with the combination of radiotherapy, fluzoparib, abiraterone acetate (II) for patients with metastatic castration-resistant prostate cancer (mCRPC).Eligible subjects who meet the inclusion criteria will be enrolled and assessed for Homologous Recombination Repair (HRR) mutation status. Participants will undergo two phases of treatment: the induction phase and the maintenance phase. During the induction phase, patients will receive Intensity-Modulated Radiation Therapy (IMRT) in combination with fluzoparib, abiraterone acetate (II), and prednisone. In the maintenance phase, patients will continue treatment with fluzoparib, abiraterone acetate (II), and prednisone. Each treatment cycle is 28 days long, and treatment will continue until disease progression is determined by the investigator and the patient is no longer clinically benefiting from the study. Follow-up will continue until the subject withdraws informed consent or the study ends, whichever occurs first.The study plans to enroll 40 eligible subjects. The primary endpoint is the PSA response rate (the proportion of patients with a ≥50% decrease in PSA from baseline). Secondary endpoints include radiographic progression-free survival (rPFS), time to PSA progression (TTPP), PSA depth of response (PSA 90, PSA undetectable rate), time to first subsequent treatment (TFST), failure-free survival (FFS), and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, male
2. ECOG score is 0 or 1
3. Untreated first-line metastatic castration resistant prostate cancer patients
4. Allow the use of a new endocrine drug treatment once during hormone sensitive stages
5. The organ function level must meet the following requirements (no blood transfusion or hematopoietic growth factor therapy received within 2 weeks before blood routine screening): ANC ≥ 1.5 × 109/L PLT≥100×109/L； • Hb≥90 g/L； • TBIL ≤ 1.5 × ULN (excluding subjects with Gilbert syndrome) • ALT and AST ≤ 2.5 × ULN; • Cr≤1.5×ULN； • LVEF≥50%； • QTcF≤450 ms。
6. If the partner is a subject with fertility, they should undergo surgical sterilization or agree to receive it during and at the end of the trial period
7. Sign a written informed consent form and expect good compliance with the research protocol

Exclusion Criteria:

1. Previously received any PARPi treatment for prostate cancer (including but not limited to Olaparib, Nilaparib, Terazopanib, Lucaparib, etc.)
2. Other clinical trial drug treatments and major surgeries received within the 4 weeks prior to randomization in this study
3. There are factors such as inability to swallow, chronic diarrhea and intestinal obstruction, or other factors that affect medication intake and absorption
4. Have a history of epilepsy or have experienced a disease that can trigger epileptic seizures within the 12 months prior to randomization (including a history of transient ischemic attacks, stroke, traumatic brain injury with consciousness disorders requiring hospitalization)
5. Active heart disease within the first 6 months of randomization, including severe/unstable angina, myocardial infarction, symptomatic congestive heart failure (heart function class III or IV), and drug-induced ventricular arrhythmias
6. Individuals with active HBV and HCV infection (HBsAg positive and virus copy number ≥ 500 IU/mL, HCV antibody positive and HCV RNA above the detection limit of the analytical method)
7. Individuals with a known history of allergies to Fluzopanib and Abiraterone nanocrystals and their components
8. Individuals with a history of congenital immunodeficiency or organ transplantation, or HIV positive subjects who meet one or more of the following criteria: Not receiving highly effective antiretroviral therapy; Change antiretroviral therapy within 6 months prior to the start of screening; • Undertaking antiretroviral therapy that may interfere with the investigational drug (please consult the sponsor before enrollment); CD4 count<350/mm3 during screening; Opportunistic infections that meet the definition of acquired immunodeficiency syndrome occurred within the 12 months prior to the start of screening
9. Patients with other malignant tumors within the past 3 years prior to randomization (excluding in situ cancer that has completely resolved and malignant tumors judged by researchers to have slow progression)
10. The researchers determined that participants with ejaculation ability and sexual activity were unwilling to take the contraceptive measures specified in the protocol during the entire study treatment period and within 3 months after the last dose

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
PSA relief rate | The duration from the first day of patient enrollment to the time when PSA decreases by ≥ 50% compared to baseline should not exceed 12 months.
  The proportion of patients who achieve a ≥50% reduction in serum PSA levels compared to baseline.

SECONDARY OUTCOMES:
Radiographic Progression-free survival（rPFS） | The duration of evaluation from the first day of patient enrollment to the time of radiological progression should not exceed 60 months.
  From the first day of patient enrollment to the time of imaging progression or death. Imaging progress includes the discovery of at least 2 new lesions under bone scanning (based on the definition of PCWG-3), or measurable soft tissue lesions under computed tomography (CT) or magnetic resonance imaging (MRI) (based on the definition of RECIST 1.1). According to the RECIST 1.1 guidelines, progression requires a 20% increase in the sum of all target lesion diameters, and an absolute minimum sum increase of 5 millimeters (mm) compared to the sum of the lowest values
Time To PSA Progression（TTPP） | The duration of evaluation from the first day of patient enrollment to the time of PSA progression should not exceed 60 months.
  To determine the progression time of prostate-specific antigen (PSA), according to the PCWG3 standard, PSA progression is defined as an increase in PSA level by ≥ 25% and an absolute value of ≥ 2µg/L (2ng/mL) compared to the lowest PSA level observed after or at baseline, and confirmed during the second consecutive test at least 3 weeks later。
PSA deep relief rate | The duration from the first day of patient enrollment to the time when PSA decreases by ≥ 90% from baseline and the lowest PSA value is ≤ 0.2ng/ml should not exceed 12 months.
  The proportion of patients who achieve a ≥90% reduction in PSA levels from baseline and have a minimum PSA value of ≤0.2 ng/ml after enrollment.
Time To First Subsequent Therapy（TFST） | The duration from the first day of patient enrollment to the start of any subsequent prostate cancer treatment should not exceed 60 months.
  The time period between the enrollment date and the date of initiation of subsequent tumor treatment.
Failure-free Survival（FFS） | The duration of evaluation from the first day of patient enrollment to any degree of disease progression should not exceed 60 months.
  From enrollment until the first occurrence of documented local or regional recurrence, distant metastasis, or death from any cause, with the earliest event taking precedence. Failure-free survival is assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.for any reason, whichever occurs first. Failure free survival evaluation based on the evaluation criteria for solid tumor treatment efficacy (RECIST V1.1)
Overall survival（OS） | The duration from the first day of patient enrollment to all-cause mortality rate should not exceed 60 months.
  Overall survival is defined as the time from the first day of enrollment to the patient's death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jianbin Bi, Doctor, Study Director — First Hospital of China Medical University
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No